CLINICAL TRIAL: NCT03954366
Title: A Phase 1, Open-label, Drug-drug-interaction Study to Determine the Effect of Rucaparib on the Pharmacokinetics of Oral Rosuvastatin (Arm A) and Oral Contraceptives (Ethinylestradiol and Levonorgestrel) (Arm B) in Patients With Advanced Solid Tumors
Brief Title: Drug-Drug Interaction Study of Rucaparib, Rosuvastatin and Oral Contraceptives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CO-338-095
Record Dates: First submitted 2019-04-02; First posted 2019-05-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Neoplasms
Keywords: rucaparib; CO-338; Clovis; Clovis Oncology; PARP Inhibitor; Drug-drug Interaction
MeSH Terms: conditions — Neoplasms | interventions — rucaparib; Rosuvastatin Calcium; Contraceptives, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - rucaparib and oral rosuvastatin (Other)
  Interventions: Drug: Rucaparib; Drug: Rosuvastatin
- Arm B - rucaparib and oral contraceptives (Other)
  Interventions: Drug: Rucaparib; Drug: Oral Contraceptives

INTERVENTIONS:
Drug: Rucaparib — Rucaparib 600 mg BID commencing on Day 5 until Day 23.
  Other Names: Rubraca
Drug: Rosuvastatin — Single dose of 20mg oral rosuvastatin on Day 1 and Day 19 only.
  Other Names: Crestor
  Arms: Arm A - rucaparib and oral rosuvastatin
Drug: Oral Contraceptives — Single dose of combined oral contraceptive (30 μg ethinylestradiol and 150 μg levonorgestrel) on Day 1 and Day 19 only.
  Arms: Arm B - rucaparib and oral contraceptives

SUMMARY:
This study will investigate the drug-drug interactions (DDIs) between rucaparib and oral rosuvastatin (Arm A), and between rucaparib and oral ethinylestradiol and levonorgestrel (Arm B), with rucaparib as a perpetrator.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, drug-drug-interaction (DDI) study in patients with advanced solid tumor. In Part I, the effects of rucaparib (600 mg twice daily [BID]) on the PK of oral rosuvastatin (Arm A) and the combined oral contraceptives (ethinylestradiol and levonorgestrel; Arm B) will be assessed.

Part I: patients will receive single oral doses of rosuvastatin or oral contraceptives (according to assigned arm) on Day 1 and Day 19. Continuous treatment with rucaparib at 600 mg BID will commence on Day 5 and continue until the end of Part I (Day 23).

Part II (optional): treatment with rucaparib in 28-day cycles may continue (at the discretion of the Investigator) until progression of disease, unacceptable toxicity, or other reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria (All patients):

* Willing to sign the ICF and to comply with the study restrictions
* Body mass index (BMI) 18.0 to 35.0 kg/m2
* Histologically or cytologically confirmed advanced solid tumor
* Patients who, in the opinion of the Investigator, could potentially benefit from treatment with rucaparib
* ECOG performance status less than or equal to 1
* Adequate organ function

Inclusion Criteria (Arm A):

- Male or female patients ≥ 18 years of age

Inclusion Criteria (Arm B):

- Female patients ≥ 18 years of age

Exclusion Criteria (All patients):

* Specific cancer treatments within 14 days prior to Day 1
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, acute coronary syndrome, cardiac angioplasty, stenting, or poorly controlled hypertension within the last 3 months prior to screening
* Pre-existing duodenal stent, recent or existing bowel obstruction
* Untreated or symptomatic central nervous system (CNS) metastases. Patients with treated asymptomatic CNS metastases are eligible
* Known HIV or AIDS-related illness, acute or history of chronic hepatitis B or C
* Female patients who are pregnant or breastfeeding
* Participation in another investigational drug trial within 30 days prior to Day 1 or exposure to more than 3 new investigational agents within 12 months prior to Day 1
* Presence of active infection requiring antibiotics
* Active second malignancy
* History of drug abuse (including alcohol)

Exclusion Criteria (Arm A):

* Current use of rosuvastatin or any other statin
* History of hypersensitivity to rosuvastatin
* Current, or history of, clinically significant myopathy

Exclusion Criteria (Arm B):

* Current use of any 1 of the contraceptive drugs or previous contraceptive implants or depot injections, which may still be clinically effective
* History of hypersensitivity to ethinylestradiol or levonorgestrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both male and female patients are eligible for Arm A. Female patients only are eligible for Arm B.
Enrollment: 36 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Maximum plasma concentration (Cmax)
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Area under the concentration-time curve (AUC) from time zero up to the last time point with a quantifiable concentration (AUC0-last)
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  AUC up to time infinity, with extrapolation of the terminal phase (AUC0-inf)

SECONDARY OUTCOMES:
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Terminal half-life (t1/2)
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Time to occurrence of Cmax (tmax)
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Apparent total clearance of drug after oral administration (CL/F)
PK parameters for oral rosuvastatin, ethinylestradiol and levonorgestrel without and with rucaparib treatment. | Day 1 to Day 23
  Apparent volume of distribution during terminal phase (Vz/F)
The following secondary PK parameter will be calculated for rucaparib. | Day 1 to Day 23
  Trough plasma concentration (Cmin)
Incidence of Adverse Events [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)
Incidence of clinical laboratory abnormalities [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)
Incidence of dose modifications [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)

CONTACTS AND LOCATIONS:
Locations (7):
- PRA Magyarország Fázis I-es Klinikai Farmakológiai Vizsgálóhely FMC Dialízis Központ, II. em., Budapest, Hungary
- Poland (5):
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej, Biała Podlaska
  - BioVirtus Centrum Medyczne, Józefów
  - Ujastek Sp. z o.o. Centrum medyczne, Krakow
  - Med Polonia Sp. z o.o., Poznan
  - Zdrowie Kobiety Centrum Leczniczo-Rehabilitacyjne i Medycyny Pracy ATTIS Sp. z o.o., Zakład Onkologii Kobiecej, Warsaw
- Summit Clinical Research s.r.o., Bratislava, Slovakia

REFERENCES:
- [Derived] Liao M, Jeziorski KG, Tomaszewska-Kiecana M, Lang I, Jasiowka M, Skarbova V, Centkowski P, Ramlau R, Gornas M, Lee J, Edwards S, Habeck J, Nash E, Grechko N, Xiao JJ. A phase 1, open-label, drug-drug interaction study of rucaparib with rosuvastatin and oral contraceptives in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2021 Nov;88(5):887-897. doi: 10.1007/s00280-021-04338-7. Epub 2021 Aug 9. PMID 34370076